CLINICAL TRIAL: NCT02217891
Title: IFACT: Incidental Findings in Advanced Cancer Therapy
Acronym: IFACT
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 14-159
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer; Colorectal Cancer; Bladder Cancer; Lung Cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Urinary Bladder Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

GROUPS / COHORTS (1):
- participants from existing MSK protocol 12-245: Participants' responses regarding the benefits and harms of incidental findings arising from tumor genomic profiling will be used to generate novel questionnaire items to assess the construct of perceived personal and clinical utility, which will be tested, along with items designed to assess knowledge about tumor genomic profiling and incidental findings.
  Part 2, the investigators will conduct 30-minute cognitive interviews to assess participants' understanding and opinions about the novel items designed to assess perceived personal and clinical utility of incidental findings and knowledge about incidental findings arising from tumor genomic profiling.
  Interventions: Behavioral: Semi-structured interview

INTERVENTIONS:
Behavioral: Semi-structured interview — Pts will participate in a 45-60-minute, one-on-one, audio-recorded interview. They will be conducted over the telephone or in person at the MSK Counseling Center. They will be conducted in accordance with a semi-structured interview guide developed by our study team of experts in clinical genetics, health psychology, & qualitative methodology. Topics to be covered in the interview include: 1) perceived potential benefits & harms of tumor genomic profiling; 2) interest in & perceived benefits & harms of incidental findings arising from tumor genomic profiling; 3) anticipated process & needs for decision-making about learning incidental findings; 4) interest in learning specific kinds of incidental findings (including those related to treatable diseases, different cancers, non-treatable diseases, & those that only have meaning for family members); 5) preferences about sharing incidental findings with other people; & 6) implications of & concerns about incidental findings for family.

SUMMARY:
The proposed study, IFACT - Incidental Findings in Advanced Cancer Therapy, will address this research gap by examining MSK patients' attitudes, preferences, and information needs regarding incidental findings arising from tumor genomic profiling.

DETAILED DESCRIPTION:
Part 1, the investigators will recruit 40 participants from those already enrolled in existing MSK IRB protocol #12-245 (PI: David Hyman, MD) including male and female patients who have been diagnosed with late-stage breast, colorectal, bladder, and lung cancer (some of the most common cancers in this study population).

Part 2, the investigators will recruit 20 participants from those who have actually received incidental germline findings from MSK IRB protocol #12-245 Consent Part C in order to cognitively test novel survey items about their knowledge and perceived utility of their incidental findings (note that the content of these items will be derived from the data collected in Part 1)

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* Patient enrolled on MSK protocol #12-245
* Living patient age 18 or older
* Patient diagnosed with breast cancer, colorectal cancer, bladder cancer, or lung cancer
* Patient residing in New York metro-area

Part 2:

* Living patient age 18 or older
* Consented to Part C of IRB#12-245 and has received results regardless if thereir was a pathogenic variant
* Patient diagnosed with cancer type approved for IRB#12-245 Part C (which are currently breast cancer, gynecological cancer, prostate cancer, and GU non-prostate cancer)breast cancer, colorectal cancer, bladder cancer, or lung cancer
* Patient residing in New York metro-area

Exclusion Criteria for Part 1 and 2:

* Non-English speakers because we do not have the resources to conduct and translate the interviews into other languages.
* Patient unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IFACT study participants will be recruited from existing MSK protocol #12-245.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
qualitive data | one time
  The study team will review and code the interview transcripts through a process of independent and collaborative thematic content analysis,(25-28) using ATLAS.ti (a qualitative data analysis software package) to facilitate the analysis process (29).

CONTACTS AND LOCATIONS:
Overall Officials: Jada Hamilton, PhD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/